CLINICAL TRIAL: NCT06692322
Title: Pharmacokinetics, Safety and Tolerability of Zongertinib Following Oral Administration in Male and Female Participants of Non-childbearing Potential With Different Degrees of Hepatic Impairment (Child-Pugh Classification A and B) Compared With Matched Male and Female Participants of Non-childbearing Potential With Normal Hepatic Function (an Open-label, Non-randomised, Single-dose, Parallel, Individual-matched Design Trial)
Brief Title: A Study to Test How Zongertinib is Taken up in the Blood of People With and Without Liver Problems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0020; U1111-1307-9446 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Liver Diseases; Healthy
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mild hepatic impairment (Child-Pugh A) (Experimental)
  Interventions: Drug: Zongertinib (BI 1810631)
- Moderate hepatic impairment (Child-Pugh B) (Experimental)
  Interventions: Drug: Zongertinib (BI 1810631)
- Normal hepatic function (Experimental)
  Interventions: Drug: Zongertinib (BI 1810631)

INTERVENTIONS:
Drug: Zongertinib (BI 1810631) — Film-coated tablet
  Other Names: BI 1810631, Hernexeos®

SUMMARY:
This study is open to adults between 18 and 80 years of age. People with a body mass index (BMI) between 18 and 42 kg/m^2 can take part. Women can only participate if they cannot get pregnant. This study includes people with mild liver problems, people with moderate liver problems, and people without liver problems as a matching control. The purpose of this study is to find out how mild and moderate liver problems affect how the body handles a medicine called zongertinib.

Participants take zongertinib once as tablets. Participants with liver problems are treated in a step-by-step approach with a few days in between for the doctors to review the data and make sure the participants can tolerate the treatment. Participants may continue their regular treatment for their liver problems during the study.

Participants are in the study for about 5 weeks. During this time, they visit the study site 4 times. This also includes an overnight stay for 6 nights. During study visits, the doctors regularly check participants' health and take note of any unwanted effects. To assess the study endpoints, the study staff regularly takes blood samples.

ELIGIBILITY:
inclusion criteria

* Male or female subjects of non-childbearing potential. Female subjects must be of non-childbearing potential either be a) postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of Follicle stimulating hormone (FSH) above 25 U/L and estradiol below 30 ng/L is confirmatory) or b) have proof of acceptable surgical sterilization. Subjects must use condom from time point of administration of trial medication until 30 days after drug administration.
* Age of 18 to 80 years (inclusive)
* Body mass index (BMI) of 18.0 to 42 kg/m^2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Male subjects with Women of child-bearing potential (WOCBP) partner must be willing to use highly effective methods of contraception (condom in combination with other methods or sexual abstinence) from time point of administration of trial medication until 30 days thereafter. These include:

  * Subject uses condoms
  * Subject is sexually abstinent
  * Subject is vasectomized (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate) and uses condom

Additionally female partners of male subjects must be willing to use any of the following criteria for a highly effective contraception from at least 30 days before the first administration of the male partner until 30 days thereafter:

* Use of intrauterine device or intrauterine hormone-releasing system by female partner plus use of condom
* Use of progestogen-only hormonal contraception by female partner that inhibits ovulation (injectables or implants) plus use of condom
* Use of combined (estrogen and progestogen containing) hormonal contraception by female partner that prevents ovulation (oral, intravaginal, or transdermal) plus use of condom
* Surgically sterilised (including hysterectomy or bilateral tubular occlusion) plus use of condom
* Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of FSH above 25 U/L and estradiol below 30 ng/L is confirmatory) plus use of condom

  * For group 1 and 2 only: Hepatic impairment classified as Child-Pugh A (score 5-6 points) or Child-Pugh B (score 7-9 points)
  * For group 1 and 2 only: Absence of clinically significant abnormalities, as based on a complete medical history including a full physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12- lead Electrocardiogram (ECG), and clinical laboratory tests at both screening and admission to trial site, with the exception of findings that in the opinion of the investigator are consistent with the participant's hepatic impairment
  * For group 1 and 2 only: Medication and/or treatment regimens must have been stable (i.e., no dose adjustments) for at least 4 weeks prior to the screening period and should be kept stable until study completion Fluctuating treatment regimens may be considered for inclusion on a case-by-case basis if the underlying disease is under control in the opinion of the investigator and must be agreed to by both the investigator and the sponsor's medical monitor Further inclusion criteria apply.

exclusion criteria

* Any finding in the medical examination (including BP, PR or ECG) assessed as clinically relevant by the investigator (apart from any non-severe hepatic impairment and associated underlying diseases)
* Severe hepatic impairment (classified as Child-Pugh C or score 10-15)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance (apart from values due to underlying disease)
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator (apart from underlying disease)
* Severe gastrointestinal, renal (Estimated glomerular filtration rate (eGFR) Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) <40 ml/min/1.73 m2 for the hepatic impaired patients and eGFR CKD-EPI <90 ml/min/1.73 m2 for matched controls), respiratory, cardiovascular, metabolic, immunological or hormonal disorders assessed as clinically relevant by the Investigator.
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, repetitive fainting spells, or repetitive blackouts Further exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to infinity (AUC0-∞) | up to 8 days
Maximum measured concentration of the analyte in plasma (Cmax) | up to 8 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- American Research Corporation at the Texas Liver Institute, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com